CLINICAL TRIAL: NCT02303561
Title: The Childhood Health and Asthma Management Program
Acronym: CHAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: American Lung Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201400235
Record Dates: First submitted 2014-11-25; First posted 2014-12-01 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Asthma; Obesity; Family; Child
MeSH Terms: conditions — Asthma; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHAMP (Experimental): Families assigned to this arm will receive tailored asthma education and behavioral skills focused on improving asthma and weight management.
  Interventions: Behavioral: CHAMP
- Health education (Active Comparator): Families assigned to this arm will receive tailored asthma education and general health education on a variety of topics.
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: CHAMP — Families assigned to this arm will receive tailored asthma education and behavioral skills focused on improving asthma and weight management.
  Arms: CHAMP
Behavioral: Health education — Families assigned to this arm will receive tailored asthma education and general health education on a variety of topics.
  Arms: Health education

SUMMARY:
Overweight and obese (OV/OB) children with asthma are at-risk for particularly poor health outcomes including poor asthma control, higher risk of asthma-related symptoms, and decreased quality of life. Weight loss reduces asthma symptoms, improves lung function, and increases quality of life among OV/OB adults with asthma. Little research has examined the impact of weight loss on asthma outcomes in OV/OB youth, and there is little research examining weight management interventions in OV/OB children with asthma. Behavioral family-based lifestyle interventions are successful in producing weight loss in children. To our knowledge, however, there has been no systematic effort to examine the impact of these interventions on weight status and asthma outcomes, nor has there been an effort to tailor these programs to the specific needs of OV/OB children with asthma.

The aims of this study are to develop and test the Childhood Health and Asthma Management Program (CHAMP), a behavioral family-based lifestyle intervention that is community-based to promote successful weight and asthma management in OV/OB children with asthma. The investigators propose to develop an intervention based on a previously developed behavioral family-based lifestyle intervention that was community-based and produced positive long term weight status changes in OV/OB children and tailor it for OV/OB children with asthma to create CHAMP. CHAMP will include asthma education and targeting unique barriers to weight management in OV/OB children with asthma. A focus group will be conducted with OV/OB children with asthma, ages 6-12, and their parent(s). Then a pilot randomized controlled trial of the CHAMP intervention with 32 OV/OB children with asthma, ages 6-12 years, and their parent(s). Families will be randomly assigned to CHAMP or a health education group. The investigators hypothesize that participants in CHAMP will have more effective weight and asthma management and child asthma outcomes compared to those in the general education group.

DETAILED DESCRIPTION:
At the first appointment the following information will be collected to determine eligibility for the research study. If participation is determined, a second visit will be scheduled at the end of the visit or the potential participant will be provided with a suggestion to speak with their primary care physician for other treatment options.

A measurement of height and weight will be taken, questionnaires regarding medical history, including asthma symptoms and control, and questionnaires about family background information (e.g., family income, size of family, employment, and marital status).

In addition, information concerning the following conditions will be collected and may exclude participation: dietary restriction or a medical condition that makes mild energy restriction or physical activity potentially dangerous, diagnosed with a major psychiatric disorder such as schizophrenia, bipolar disorder or autism, has used systemic corticosteroids within 3 months, or prescription weight loss drugs within 6 months.

The second appointment will happen one to two weeks before the start of the treatment program. During this visit the following will happen:

A measurement of height and weight, and waistline, questionnaires and complete an interview about asthma management and quality of life, and a test for lung function both pre and post albuterol. At the end of the visit an accelerometer will be provided to wear for 7 days in a row. The accelerometer will measure how much exercise is done each day.

At the end of this visit, the participant will be randomly assignment to either the experimental Childhood Health and Asthma Management Program (CHAMP) group or the health education group.

The CHAMP group will receive tailored asthma education and behavioral skills focused on improving asthma and weight management.

The health education group will receive tailored asthma education and general health education on a variety of topics.

Each of the treatment programs will last for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* speaks English;
* has a physician-verified persistent asthma diagnosis or by indicating on a screening questionnaire that they

  1. having a current prescription for a controller medication (e.g. Fluticasone), or
  2. demonstrating any of the following symptom frequency in the previous month: (I) daytime asthma symptoms more than two days a week, (II) nighttime awakenings due to asthma more than times a month, (III) short-acting beta agonist use 2 days a week, (IV) normal activity limitation, (V) oral steroid use 2 times a year, (VI) emergency department visit due to asthma in past year;
* has a BMI at or above the 85th percentile for age and gender norms as published by the CDC.

Participating parents of legal guardians must:

* live in the same home with the child;
* speak English;
* be aged 75 or younger. There is no BMI requirement for participating parents/legal guardians.

Exclusion Criteria:

* child or parent has dietary restriction or a medical condition that contraindicates mild energy restriction or physical activity (history of musculo-skeletal condition that limits walking, heart condition, chronic lung diseases limiting physical activity, current participation in commercial weight loss program);
* use of antipsychotic agents, monoamine oxidase inhibitors, systemic corticosteroids within 3 months, or prescription weight loss drugs within 6 months.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-13 (Actual)

PRIMARY OUTCOMES:
Spirometry will be used to test the change in lung function from baseline, 4 months, and 10 months | Change from Baseline, 4 months, and 10 months

SECONDARY OUTCOMES:
Body Mass Index will be calculated to test the change in weight from baseline, 4 months, and 10 months | Change from Baseline, 4 months, and 10 months
The Asthma Control Test questionnaire will be calculated to test the change in asthma control from baseline, 4 months, and 10 months | Change from Baseline, 4 months, and 10 months
The Family Asthma Management System Scale semi-structured interview will be used to test the change in family asthma management from baseline, 4 months, and 10 months. | Change from Baseline, 4 months, and 10 months
The Standardised Paediatric Asthma Quality of Life Questionnaire interview will be used to test the change in quality of life from baseline, 4 months, and 10 months. | Change from Baseline, 4 months, and 10 months
The Block Foods questionnaire will be used to test the change in dietary intake from baseline, 4 months, and 10 months. | Change from Baseline, 4 months, and 10 months
Objectively monitored physical activity will be used to test the change in physical activity from baseline, 4 months, and 10 months. | Change from Baseline, 4 months, and 10 months

CONTACTS AND LOCATIONS:
Overall Officials: David A Fedele, Ph.D>, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided